CLINICAL TRIAL: NCT00153751
Title: Clinical Study to Test the Efficacy of Herbal Medicine in Relieving Symptoms and Change of Quality of Life of Patients With IBS
Brief Title: The Efficacy of Herbal Medicine in Relieving Symptoms and Change of Quality of Life of Patients With Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Dr WK Leung, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JC_IBS
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-05-13 (Estimated); Status verified 2008-05

CONDITIONS: Colonic Diseases, Functional
Keywords: Traditional Chinese Medicine
MeSH Terms: conditions — Colonic Diseases, Functional | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Traditional Chinese Medicine (Experimental): They are Common peony root, other herbs.
  Interventions: Drug: Traditional Chinese Medicine
- Holopon (Active Comparator): Holopon
  Interventions: Drug: Holopon
- placebo (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Traditional Chinese Medicine — They are Common peony root, Rhizoma Atractylodis Macrocephalae, Radix Paeoniae Lactiflorae, Cortex Magnoliae Officinalis, Rhizoma Curcumae Longae, Fructus Schisandrae Chinensis, Pericarpium Citri Reticulatae, and Rhizoma Corydalis Yanhusuo.
  Other Names: TCM
  Arms: Traditional Chinese Medicine
Drug: Holopon — holopon
  Other Names: Western Medicine
  Arms: Holopon
Other: placebo — placebo
  Other Names: dummy
  Arms: placebo

SUMMARY:
To test the efficacy of herbal medicine in relieving symptoms and change of quality of life of patients with IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a diagnosis in Western Medicine characterized by recurrent abdominal pain associated with disturbance in bowel habit such as diarrhea or constipation. Epidemiological studies showed that 14% of males and 27% of females in the US (white) have symptoms of IBS. In Hong Kong, our survey reported a similar prevalence of this condition among Chinese (13% in males and 21% in females). IBS is one of the most common conditions leading to seeking of medical care. Treatment for IBS has so far been unsatisfactory. Numerous medications have been proposed for IBS; however, none is convincingly effective. A review and critique of published drug trials for IBS from 1966 to 1988 concluded that there was no proof that any western medicine is effective for all IBS patients. With the unsatisfactory treatment response of western medicine, many turned to alternative treatment modalities for IBS. Traditional Chinese medicine is particularly attractive as their effectiveness in treating functional disorders and retaining balance of body functions has been known for centuries. However, there is a lack of convincing clinical data demonstrating the effectiveness of Chinese medicine in this condition. In this study, we sought to determine the efficacy of herbal medicine in relieving symptoms and quality of life of patients with IBS. This is a prospective randomized, double-blinded double placebo-controlled study in patients with non-constipation type IBS. Patients will be randomized to receive either one of three treatment arms: 1. herbal medicine (HM) + placebo western medicine (WM), 2. WM + placebo HM and 3. placebo HM + placebo WH. Each patient will go through an 8-week period of randomized double-blind treatment with either HW, WM or placebo and followed by an 8-week of observation period. The IBS symptom and quality of life will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients (aged 18-65) attending the Gastroenterology Clinic of the Prince of Wales Hospital or Hong Kong Baptist University Chinese Medicine clinics for symptoms of IBS will be enrolled in the study.
* IBS is diagnosed by Rome II criteria [Thompson et al. Gut 2000]: At least 12 weeks, which need not be consecutive, in the preceding 12 months of abdominal discomfort or pain that has two of three features: relieved with defecation; and/or onset associated with a change in frequency of stool; and/or onset associated with a change in form (appearance) of stool
* Normal colonic evaluation (colonoscopy or barium enema) in recent 5 years
* Mean score of abdominal discomfort/pain,based on a 5-point scale,at baseline and during the 2-week run-in period
* Informed written consent for participation into study.
* Ethical approval will be obtained from the Clinical Research Ethics Committee of the University

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The global assessment of IBS symptom by patients. | 16 weeks

SECONDARY OUTCOMES:
Individual IBS symptoms and QOL assessment | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, MD, Principal Investigator — CUHK
Locations (1):
- Li Ka Shing Specialist Clinic, Prince of Wales Hospital, Hong Kong (sar), China